CLINICAL TRIAL: NCT07256418
Title: Transcriptomic Study of Cutaneous Fibroblasts in Scleroderma
Acronym: TRANSCLERO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BONNOTTE 2025-2
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scleroderma: People with systemic scleroderma
  Interventions: Procedure: Skin samples; Other: Analysis of fibroblasts
- Control: People undergoing plastic, cosmetic and reconstructive surgery
  Interventions: Procedure: Skin samples; Other: Analysis of fibroblasts

INTERVENTIONS:
Procedure: Skin samples — * Scleroderma group: skin biopsy for scleroderma patients
  * Control group: recovery of resected tissue from patients undergoing plastic, reconstructive and aesthetic surgery.
Other: Analysis of fibroblasts — Analysis of samples by RNA sequencing

SUMMARY:
Scleroderma is a complex connective tissue disease involving three interconnected pathophysiological axes: vascular hyperactivity and remodelling, immune system dysfunction and over-activation of fibroblasts at the origin of the fibrosis process in the skin and organs. Given that this pathology occurs preferentially in mature subjects, it is possible to suggest a potential inductive role for senescent fibroblasts, which would be responsible for activating and/or maintaining the immune response and systemic inflammation. Our hypothesis is that fibroblasts play a predominant role in the genesis and maintenance of this pathology.

ELIGIBILITY:
Inclusion Criteria:

FOR PATIENTS WITH SCLERODERMA :

* Person who has given written consent
* Person with systemic scleroderma

FOR CONTROL PARTICIPANTS :

* Person who has given written consent
* Person undergoing plastic, cosmetic and reconstructive surgery

Exclusion Criteria:

FOR PATIENTS WITH SCLERODERMA :

* Person not affiliated to or not benefiting from a social security scheme
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* An adult who is incapable or unable to give consent
* Minors

FOR CONTROLLED PARTICIPANTS :

* Person suffering from a chronic disease or under chronic treatment for autoimmune, inflammatory or dermatological diseases
* Person not affiliated to or not benefiting from a social security scheme
* Person under legal protection (curatorship, guardianship)
* Person subject to a legal protection measure
* An adult who is incapable or unable to give consent
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants (patients and control participants) will be identified during their usual follow-up consultation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
genes involved in the various cell activation and signalling pathways | through study completion, an average of 12 months
  number and type of genes involved in different cell activation and signalling pathways, including senescence, which will be differentially expressed in fibroblasts from the skin of control participants and those from the skin of subjects with SSc.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France